CLINICAL TRIAL: NCT01588678
Title: A Phase 1, Open-Label, Multiple Ascending Dose Study of DS-3078a, an Oral TORC1/2 Kinase Inhibitor, in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: A Open-Label, Multiple Ascending Dose Study of DS-3078a, an Oral TORC1/2 Kinase Inhibitor, in Subjects With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS3078-A-U101
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2015-04

CONDITIONS: Advanced Solid Tumor; Lymphoma
Keywords: endometrial; prostate; breast; gastric; cervical; ovarian; neuroendocrine cancers; soft-tissue sarcoma; squamous cell NSCLC; renal cell carcinoma; non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Sarcoma; Carcinoma, Renal Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS-3078a (Experimental): Part 1 - Dose escalation of DS-3078a to determine the maximum tolerated dose (MTD) will be guided by the modified continuous reassessment method (mCRM) using a Bayesian logistic regression model (BLRM) following escalation with overdose control (EWOC) principle.
  Before starting mCRM, initial dose escalation will proceed following an accelerated titration in which single subjects will be enrolled into sequential dose levels with a dose increment of up to 100% from the previous dose.
  Upon completion of Part 1 with established MTD and tentative recommended phase 2 dose (RP2D), the Dose Expansion (Part 2) will begin with the intention of further assessing the safety and tolerability of DS-3078a, confirming the RP2D, determining the Pharmacodynamic response in tumor samples, and evaluating preliminary efficacy of DS-3078a in subjects.
  Interventions: Drug: DS-3078a

INTERVENTIONS:
Drug: DS-3078a — DS-3078a will be administered as oral capsules once daily and will be supplied in 5, 20, 50, and 150 mg capsules.

SUMMARY:
DS-3078a will be evaluated as a single agent in subjects with advanced solid tumor malignancies or lymphomas refractory to standard treatment or for which no standard treatment is available.

DETAILED DESCRIPTION:
This is a Phase 1, open-label study of DS-3078a to assess safety and tolerability, identify the maximum tolerated dose (MTD) and tentative recommended phase 2 dose (RP2D), and assess pharmacokinetic and pharmacodynamic properties in subjects with advanced solid tumor malignancies or lymphomas. The study will include 2 parts: Dose Escalation and Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* A pathologically or cytologically documented advanced solid tumor or lymphoma that has relapsed from or is refractory to standard treatment or for which no standard treatment is available.
* Men or women >=18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status =<1
* Have adequate bone marrow function, defined as:

  * Platelet count >=100 x 10^9/L for solid tumors and >=75 x 10^9/L for lymphomas,
  * Hemoglobin level >=9.0 g/dL, and ANC >=1.5 x 10^9/L for solid tumors and >=1.0 x 10^9/L for lymphomas.
* Have adequate renal function, defined as:

Creatinine clearance >=60 mL/min, or creatinine =<1.5 x ULN.

* Have adequate hepatic function, defined as:

  * AST/ALT levels =<3 x ULN (=<5 x ULN if liver metastases are present) and
  * Bilirubin =<1.5 x ULN.
* Have adequate blood clotting function, defined as prothrombin time and activated partial thromboplastin time =<1.5 x ULN.
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Institutional Review Board/Ethics Committee-approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study specific procedures or tests.

For Part 2

* A pathologically or cytologically documented advanced solid tumor or non-Hodgkin lymphoma, with measurable disease based on RECIST 1.1 or revised IWG criteria, that is refractory to standard treatment. The solid tumor types that will be included in the study are of the following kinds in which the mTOR signaling is frequently activated: endometrial, prostate, breast, gastric, cervical,ovarian, or neuroendocrine cancers, soft-tissue sarcoma, squamous cell NSCLC,renal cell carcinoma or other tumor types approved by the Sponsor.
* Agree to undergo pre- and post-treatment tumor biopsies.

Exclusion Criteria:

* History of primary central nervous system malignancies
* Gastrointestinal diseases that could affect the absorption of DS-3078a in the opinion of the Investigator
* Subjects with a fasting glucose >126 mg/dL (>7 mmol/L)
* History of diabetes mellitus (type 1 or 2) or glycosylated hemoglobin >7.0% at screening
* Positive test for hepatitis B surface antigen or hepatitis C antibody
* Recipient of live vaccine within 1 month of or during study drug treatment
* Use of chronic systemic corticosteroids (use of nasal or inhaled steroids is permitted)
* Subjects requiring daily supplemental oxygen
* Recipient of an allogenic stem cell or bone marrow transplant
* Presence of a concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor
* Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE v4 grade =<1 or baseline.
* Systemic treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy within 3 weeks before study drug treatment; or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment; or treatment with small-molecule targeted agents within 2 weeks or 5 half-lives before study drug treatment, whichever is longer.
* Therapeutic radiation or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment
* Participation in a clinical study within 3 weeks (2 weeks or 5 half-lives, whichever is longer, for small-molecule targeted agents) before study drug treatment, or current participation in other investigational procedures
* Concomitant treatment with strong inhibitors or inducers of cytochrome P450 3A4 and P glycoprotein
* Less than 1 week since using systemically acting drugs that increase gastric pH, such as H2-blockers and proton pump inhibitors. Antacids should be avoided within 48 hours of the first dose of DS 3078a
* Prolongation of corrected QT interval by Fridericia's method (QTcF) at rest, where the mean QTcF interval is >450 msec based on triplicate electrocardiogram (ECG)
* Pregnant or breastfeeding
* Substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results

For Part 2

* Subjects who have had prior treatment with an mTOR catalytic site inhibitor or dual PI3K/mTOR inhibitor (including, but not limited to, OSI-027, INK128, ADZ8055,AZD2014, WYE12513, PP242, BEZ-235, DS-7423, XL765, GDC-0980, SF1126, GSK2126458, PF4691502, and PF05212384) will be disqualified from entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 3 years
  To determine the maximum tolerated dose (MTD) and tentative recommended Phase 2 dose (RP2D) of DS 3078a

SECONDARY OUTCOMES:
determine the Cmax profile of DS 3078a | 3 years
  determine the Cmax (maximum concentration) of DS-3078a administered under fed and unfed conditions
effect on glucose metabolism | 3 years
  determine the effect of DS-3078a on glucose metabolism by measuring serum glucose and C peptide
assess pharmacodynamic effects tumor glucose uptake | 3 years
  assess the pharmacodynamic effects of DS 3078a by determining tumor glucose uptake using (18F) fluorodeoxyglucose positron emission tomography (FDG-PET)
assess tumor response | 3 years
  assess tumor response to DS-3078a in subjects with advanced non-Hodgkin lymphomas or advanced solid tumor types in which the mammalian target of rapamycin (mTOR) signaling pathway is frequently activated
assess pharmacodynamic effects v-akt murine thymoma viral oncogene | 3 years
  assess the pharmacodynamic effects of DS 3078a by measuring v-akt murine thymoma viral oncogene homolog 1 (Akt) phosphorylation in platelet rich plasma (PRP)
determine the AUC of DS 3078a | 3 years
  determine the Area under the concentration versus time curve (AUC) of DS-3078a administered under fed and unfed conditions
determine the Tmax of DS 3078a | 3 years
  determine the time of maximum concentyration (Tmax) of DS-3078a administered under fed and unfed conditions
determine the terminal half-life of DS 3078a | 3 years
  determine the terminal half-life (T1/2) of DS-3078a administered under fed and unfed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- South Texas Accelerated Research Therapeutics, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/